CLINICAL TRIAL: NCT06448897
Title: Development of an Imaging Prediction Model for Pelvic Lymph Node Metastasis of Cervical Cancer Using Artificial Intelligence Techniques.
Status: Recruiting | Type: Observational
Sponsor: Obstetrics & Gynecology Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: FUOBGY2024-33
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Cervical Cancer; Lymph Node Metastasis; Artificial Intelligence
Keywords: Cervical Cancer; Lymph Node Metastasis; Artificial Interlligence
MeSH Terms: conditions — Uterine Cervical Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a retrospective exploratory trial conducted at a single center, aiming to develop and validate a preoperative lymphatic metastasis model for cervical cancer using artificial intelligence deep learning. The model is trained using preoperative imaging and postoperative pathological findings of cervical cancer patients, with the goal of enhancing the accuracy of lymphatic metastasis prediction through preoperative imaging and offering insights for treatment decisions.

ELIGIBILITY:
Inclusion criteria:

1. patients with preoperative diagnosis of invasive cervical cancer stage I-III, with any type of pathology, and patients who underwent radical/modified radical cervical cancer surgery + pelvic lymph node dissection in our hospital.
2. Age ≥18 years old and ≤80 years old
3. patients with complete preoperative pelvic MRI images and postoperative pathology and clinical data in our hospital

Exclusion criteria:

1. Patients during pregnancy or breastfeeding, patients within 42 days of abortion
2. Patients who have received neoadjuvant chemotherapy or radiotherapy before surgery for this previous cervical cancer
3. Patients with other malignant tumors within 5 years
4. Combination of other underlying diseases that may lead to enlarged pelvic lymph nodes
5. Imaging report more than 1 month prior to surgery
6. Poor image quality and unrecognizable

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patient information and imaging data were collected from the Obstetrics and Gynecology Hospital of Fudan University. This hospital is a specialized tertiary care facility and is recognized as the leading Obstetrics and Gynecology hospital in China.
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
A model for identifying pelvic lymph node metastases on preoperative imaging | From enrollment to the end of development of model at 24 months
  Artificial intelligence (AI) technology was utilized to develop a model for identifying pelvic lymph node metastasis from preoperative images in order to enhance the accuracy of preoperative lymph node metastasis detection in cervical cancer. The model was validated with the main diagnostic focus on determining the status of lymph node metastasis.

CONTACTS AND LOCATIONS:
Locations (1):
- The Obstetrics and Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No